CLINICAL TRIAL: NCT04018131
Title: The Efficacy of Cimetidin for Acute - Extrinsic Atopic Dermatitis Treated With Standard Therapy, a Study of Immunoglobulin E, Interleukin-4, Interleukin-12, and Interferon-Ɣ Serum Levels
Brief Title: The Efficacy of Cimetidin for Acute - Extrinsic Atopic Dermatitis Treated With Standard Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0071
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Atopic Dermatitis; Immunoglobulin E Concentration, Serum
Keywords: Atopic Dermatitis; Cimetidine; Immunoglobulin E; Interleukin-4; Interleukin-12; Interferon Gamma; SCORAD; Treatment
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Cimetidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cimetidine (Active Comparator)
  Interventions: Drug: Cimetidine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Cimetidine — Antihistamine 2 antagonist
  Arms: Cimetidine
Drug: Placebos — Placebo drug
  Arms: Placebo

SUMMARY:
Extrinsic - atopic dermatitis is characterized by increased of IgE serum levels. Acute extrinsic - atopic dermatitis is a type 1 hypersensitivity that involve various inflammatory mediator including Interleukin-4, Interleukin-12, and Interferon-Ɣ. Recent treatment of atopic dermatitis mainly focused on reducing the inflammation through topical and systemic regiments. However, no systemic medication could control the atopic dermatitis remission yet, and the current immunosuppressive agent used may cause many side effects if administered on a long term basis.

In the future, treatment of atopic dermatitis were specifically targeted to inhibit the role of Th2. Cimetidine is H2 receptor antihistamine that has been widely used as gastrointestinal medication for a long time. Cimetidine could modulate the immune system by activating the Th1 and lowering the Th2 activity, and lowering the IgE levels thus reducing the severity of atopic dermatitis.

DETAILED DESCRIPTION:
The aim of this study is to measure the efficacy of cimetidine for acute, extrinsic-atopic dermatitis treated with standard therapy using SCORAD as the clinical outcome. This study also measure Immunoglobulin E, Interleukin-4, Interleukin-12, and Interferon-Ɣ serum levels before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Atopic dermatitis patients diagnosed with Hanifin Rajka criteria
* Acute extrinsic atopic dermatitis
* IgE levels above 200 IU/mL
* Minimum weight 15kg

Exclusion Criteria:

* Consumption of corticosteroid and systemic immunosuppressant within the last 2 weeks
* Chronic lesion
* Consumption of drugs that reacts with cimetidine
* Disturbance in lab results including complete blood count, liver function, and renal function.
* Other conditions that might increase IgE levels

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2018-03-26 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
SCORAD change | 0, 2, 4, 6, 8 weeks
  Scoring Atopic Dermatitis (SCORAD) is a score to indicate the severity of atopic dermatitis.
  The minimum score is 0, maximum score is 103. Mild 0 - 14 Moderate 15 - 39 Severe 40 - 103
  The SCORAD before treatment was expected to be higher than after treatment. Outcome: change of SCORAD
Immunoglobulin E change | 0, 8 weeks
  Change of Immunoglobulin E

SECONDARY OUTCOMES:
Interleukin-4 change | 0, 8 weeks
  Change of Interleukin-4
Interleukin-12 change | 0, 8 weeks
  Change of Interleukin-12
Interferon Gamma change | 0, 8 weeks
  Change of Interferon Gamma

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Novianto E, Jacoeb TNA, Indriatmi W, Suhendro, Setiabudy R, Setiabudy RD, Abdullah M, Rengganis I, Suwarsa O, Soebaryo RW. Effectiveness of Cimetidine as Adjuvant Therapy in the Treatment of Acute-Extrinsic Atopic Dermatitis: A Double-Blind Randomized Controlled Trial. Dermatol Ther (Heidelb). 2022 Mar;12(3):715-726. doi: 10.1007/s13555-022-00688-z. Epub 2022 Feb 17. PMID 35175572